CLINICAL TRIAL: NCT01467882
Title: An Open-label, Non-comparative, Multicenter Study on the Efficacy, Safety, and Pharmacokinetics of Triptorelin Pamoate (Embonate) 22.5 mg 6-month Formulation in Patients Suffering From Central (Gonadotropin-dependent) Precocious Puberty
Brief Title: Efficacy, Safety, and Pharmacokinetics (PK) of Triptorelin 6-month Formulation in Patients With Central Precocious Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 8206-CPP-301
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2015-09-04 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triptorelin (Experimental): Triptorelin 22.5 mg, intramuscular (IM), at Day 1 and Day 169
  Interventions: Drug: Triptorelin

INTERVENTIONS:
Drug: Triptorelin — Powder and solution for solution for injection
  Other Names: Trelstar

SUMMARY:
The study will investigate the efficacy, safety and pharmacokinetics of triptorelin 22.5 mg 6-month formulation in 44 patients suffering from central precocious puberty. The total study duration per patient will be 12 months (48 weeks).

ELIGIBILITY:
Inclusion criteria:

1. Onset of development of sex characteristics before 8 and 9 years in girls and boys, respectively (breast development in girls or testicular enlargement in boys according to the Tanner method), and candidate to receive at least 12 months of GnRH agonist therapy after study entry.
2. Aged 2-8 years inclusive (i.e. < 9 years) for girls and 2-9 years inclusive (i.e. < 10 years) for boys at initiation of triptorelin treatment.
3. Initiation of triptorelin treatment at the latest 18 months after onset of the first signs of precocious puberty.
4. Difference (Δ) bone age (Greulich and Pyle method) - chronological age ≥ 1 year.
5. Pubertal-type LH response 30 minutes following a GnRH agonist stimulation test before treatment initiation (leuprolide acetate 20 μg/kg SC) ≥ 6 IU/L.
6. Clinical evidence of puberty, defined as Tanner Staging ≥ 2 for breast development for girls and testicular volume ≥ 4 mL (cc) for boys.
7. Informed consent signed by one parent or both parents (as per local requirements), by the liable parent or by the legal guardian (when applicable); assent signed by the child if ≥ 7 years.

Non-inclusion criteria:

1. Gonadotropin-independent (peripheral) precocious puberty: extra pituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroid secretion.
2. Non-progressing isolated premature thelarche.
3. Presence of an unstable intracranial tumour or an intracranial tumour requiring neurosurgery or cerebral irradiation. Patients with hamartomas not requiring surgery are eligible.
4. Evidence of renal (creatinine > 2 x ULN) or hepatic impairment (bilirubin or ASAT > 3 x ULN).
5. Any other condition or chronic illness or treatment possibly interfering with growth or other study endpoints (e.g. chronic steroid use [except mild topical steroids], renal failure, diabetes, moderate to severe scoliosis, previously treated intracranial tumour).
6. Prior or current therapy with a GnRH agonist, medroxyprogesterone acetate, growth hormone or insulin-like growth factor-1 (IGF 1).
7. Major medical or psychiatric illness that could interfere with study visits.
8. Diagnosis of short stature, i.e. > 2.25 SD below the mean height for age.
9. Positive pregnancy test.
10. Known hypersensibility to any of the test materials or related compounds.
11. Use of anticoagulants (heparin and coumarin derivatives).

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tala Dajani, MD, Principal Investigator — Pediatric Endocrinology of Phoenix, Arizona; Barry Reiner, MD, Principal Investigator — Barry J. Reiner, MD, LLC, Baltimore, Maryland; Galal Salem, MD, Principal Investigator — SRCR, Inc, Bell Gardens, California; Heidi Shea, MD, Principal Investigator — Endocrine Associates of Dallas, Plano, Texas; Mark Rappaport, MD, Principal Investigator — Pediatric Endocrine Associates, Atlanta, Georgia; Opada Alzohaili, MD, Principal Investigator — Alzohaili Medical Consultants, Dearborn, Michigan; Quentin Van Meter, MD, Principal Investigator — Van Meter Pediatric Endocrinology, Peachtree City, Georgia; David Domek, MD, Principal Investigator — Lynn health Science Institute, Oklahoma City; Kathleen Bethin, MD, Principal Investigator — Women's & Children's Hospital of Buffalo, New York; Paul Kaplowitz, MD, Principal Investigator — Children's National Medical Center, Washington; Karen Klein, MD, Principal Investigator — Children's National Medical Center, San Diego, California; Diane Merritt, MD, Principal Investigator — Washington University, St. Louis, Missouri; Susan Rose, MD, Principal Investigator — Cincinnati Children's Hospital, Ohio; Gad Kletter, MD, Principal Investigator — Swedish Pediatric Specialist, Seattle, Washington; Javier Aisenberg, MD, Principal Investigator — Hackensack university medical center, New Jersey; Dennis Brenner, MD, Principal Investigator — St. Barnabas Medical Center, Livingston, New Jersey; Douglas Rogers, MD, Principal Investigator — Cleveland Clinic, Ohio; Lawrence Silverman, MD, Principal Investigator — Goryeb Children's Hospital, Morristown, New Jersey; Peter Lee, MD, Principal Investigator — Penn State Hershey Children's Hospital, Pennsylvania; Ricardo Gomez, MD, Principal Investigator — Children's Hospital, New Orleans, Louisiana; Fernando Cassorla, MD, Principal Investigator — IDIMI, Santiago, Chile; Joshua Yang, MD, Principal Investigator — Arnold Palmer Pediatric Endocrinology Practice, Orlando, Florida; Erica Eugster, MD, Principal Investigator — James Whitcomb Riley Hospital for Children, Indianapolis, Indiana; Oscar Flores, MD, Principal Investigator — Hospital Universitario de Monterrey, Mexico; Nancy Wright, MD, Principal Investigator — Nancy Wright MD P.A., Tallahasse, Florida
Locations (13):
- United States (11):
  - Pediatric Endocrinology of Phoenix, Phoenix, Arizona
  - Children's National Medical Center, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Arnold Palmer Pediatric Endocrinology Practice, Orlando, Florida
  - Nancy Wright MD P.A., Tallahassee, Florida
  - Washington University, St Louis, Missouri
  - Hackensack university medical center, Hackensack, New Jersey
  - Women's & Children's Hospital of Buffalo, Buffalo, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Lynn health Science Institute, Oklahoma City, Oklahoma
  - Swedish Pediatric Specialist, Seattle, Washington
- IDIMI, Santiago, Chile
- Hospital Universitario de Monterrey, Monterrey, Mexico

REFERENCES:
- [Background] Carel JC, Eugster EA, Rogol A, Ghizzoni L, Palmert MR; ESPE-LWPES GnRH Analogs Consensus Conference Group; Antoniazzi F, Berenbaum S, Bourguignon JP, Chrousos GP, Coste J, Deal S, de Vries L, Foster C, Heger S, Holland J, Jahnukainen K, Juul A, Kaplowitz P, Lahlou N, Lee MM, Lee P, Merke DP, Neely EK, Oostdijk W, Phillip M, Rosenfield RL, Shulman D, Styne D, Tauber M, Wit JM. Consensus statement on the use of gonadotropin-releasing hormone analogs in children. Pediatrics. 2009 Apr;123(4):e752-62. doi: 10.1542/peds.2008-1783. Epub 2009 Mar 30. PMID 19332438
- [Background] Martinez-Aguayo A, Hernandez MI, Beas F, Iniguez G, Avila A, Sovino H, Bravo E, Cassorla F. Treatment of central precocious puberty with triptorelin 11.25 mg depot formulation. J Pediatr Endocrinol Metab. 2006 Aug;19(8):963-70. doi: 10.1515/jpem.2006.19.8.963. PMID 16995580
- [Background] Houk CP, Kunselman AR, Lee PA. The diagnostic value of a brief GnRH analogue stimulation test in girls with central precocious puberty: a single 30-minute post-stimulation LH sample is adequate. J Pediatr Endocrinol Metab. 2008 Dec;21(12):1113-8. doi: 10.1515/jpem.2008.21.12.1113. PMID 19189683
- [Background] Lahlou N, Carel JC, Chaussain JL, Roger M. Pharmacokinetics and pharmacodynamics of GnRH agonists: clinical implications in pediatrics. J Pediatr Endocrinol Metab. 2000 Jul;13 Suppl 1:723-37. doi: 10.1515/jpem.2000.13.s1.723. PMID 10969915
- See also: Study sponsor — http://www.debiopharm.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Intention to treat, defined as all participants enrolled
Groups:
- Children: All children enrolled who received triptorelin 22.5 mg, intramuscular (IM), at Day 1 and Day 169
Period: Overall Study
Arm/Group | Children
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat, defined as all participants enrolled
Arm/Group | Children
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.41 (1.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 28
  Mexico | 1
  Chile | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Children With Luteinizing Hormone (LH) Suppression to Prepubertal Levels 30 Minutes After Leuprolide Stimulation at Month 6
Description: This is a lab test to see what percentage of participants were returned to normal before-puberty levels at Month 6.
Time Frame: Month 6
Population: Intention to treat, defined as all participants enrolled
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants | 93.18 [81.34 to 98.57]

2. Secondary Outcome: Percentage of Children With LH Suppression to Prepubertal Levels 30 Minutes After Leuprolide Stimulation at Months 1, 2, 3, 9 and 12
Description: This is a lab test to see what percentage of children were returned to normal before-puberty levels by the drug at each time point.
Time Frame: at Months 1, 2, 3, 9 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants
  Month 1 | 95.45
  Month 2 | 95.45
  Month 3 | 95.45
  Month 9 | 95.45
  Month 12 | 97.73

3. Secondary Outcome: Percentage of Children Maintaining LH Suppression at Prepubertal Levels 30 Minutes After Leuprolide Stimulation From Month 6 to 12
Description: This is a lab test to see what percentage of children stayed at the normal before-puberty level from month 6 to month 12.
Time Frame: from Month 6 to 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants | 93.18

4. Secondary Outcome: Percentage of Children With LH Suppression (LH ≤ 4 IU/L)30 Minutes After Leuprolide Stimulation at Months 1, 2, 3, 6, 9 and 12
Description: This is a lab test to see what percentage of children were returned to lower than normal before-puberty levels by the drug at each time point.
Time Frame: at Months 1, 2, 3, 6, 9 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants
  Month 1 | 95.45
  Month 2 | 95.45
  Month 3 | 93.18
  Month 6 | 90.91
  Month 9 | 93.18
  Month 12 | 97.73

5. Secondary Outcome: Percentage of Children Maintaining LH Suppression at </= 4 IU/L 30 Minutes After Leuprolide Stimulation From Month 6 to 12
Description: This is a lab test to see what percentage of children stayed at the lower than normal before-puberty level from month 6 to month 12.
Time Frame: from Month 6 to 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants | 90.91

6. Secondary Outcome: Change From Baseline in Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) at Months 1, 2, 3, 6, 9, and 12
Time Frame: Baseline to Months 1, 2, 3, 6, 9, and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Mean (Standard Deviation); unit: IU/L
Groups:
- All Children Luteinizing Hormone; All Children Follicle Stimulating Hormone: All children enrolled who received triptorelin 22.5 mg, intramuscular (IM), at Day 1 and Day 169
Arm/Group | All Children Luteinizing Hormone | All Children Follicle Stimulating Hormone
Number analyzed (Participants) | 44 | 44
IU/L
  at Month 1 | -25.21 (20.28) | -8.85 (4.15)
  at Month 2 | -25.25 (20.41) | -8.80 (4.20)
  at Month 3 | -25.17 (20.53) | -8.13 (4.26)
  at Month 6 | -23.06 (22.17) | -6.66 (4.61)
  at Month 9 | -25.24 (20.49) | -7.87 (4.27)
  at Month 12 | -25.15 (20.50) | -6.99 (4.63)

7. Secondary Outcome: Change From Baseline in Estradiol Levels at Months 1, 2, 3, 6, 9, and 12
Time Frame: Baseline to Months 1, 2, 3, 6, 9, and 12
Population: Intention to treat girls, defined as all girls enrolled
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- Girls: All girls enrolled who received triptorelin 22.5 mg, intramuscular (IM), at Day 1 and Day 169
Arm/Group | Girls
Number analyzed (Participants) | 39
ng/L
  at Month 1 | -31.87 (27.82)
  at Month 2 | -31.24 (31.80)
  at Month 3 | -32.15 (28.65)
  at Month 6 | -28.18 (31.26)
  at Month 9 | -30.08 (27.44)
  at Month 12 | -29.74 (28.24)

8. Secondary Outcome: Change From Baseline in Testosterone Levels at Months 1, 2, 3, 6, 9, and 12
Time Frame: Baseline to Months 1, 2, 3, 6, 9, and 12
Population: Intention to treat boys, defined as all boys enrolled
Measure: Mean (Standard Deviation); unit: ng/dL
Groups:
- Boys: All boys enrolled who received triptorelin 22.5 mg, intramuscular (IM), at Day 1 and Day 169
Arm/Group | Boys
Number analyzed (Participants) | 5
ng/dL
  at Month 1 | -306.96 (184.06)
  at Month 2 | -290.70 (214.81)
  at Month 3 | -319.20 (177.04)
  at Month 6 | -317.62 (178.11)
  at Month 9 | -315.54 (183.98)
  at Month 12 | -301.86 (205.29)

9. Secondary Outcome: Percentage of Children With Prepubertal Estradiol or Testosterone Levels at Months 1, 2, 3, 6, 9, and 12
Time Frame: at Months 1, 2, 3, 6, 9, and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children | Girls | Boys
Number analyzed (Participants) | 44 | 39 | 5
percentage of participants
  at Month 1 | 86.36 | 87.18 | 80.00
  at Month 2 | 88.37 | 89.47 | 80.00
  at Month 3 | 93.18 | 92.31 | 100.00
  at Month 6 | 81.82 | 79.49 | 100.00
  at Month 9 | 81.82 | 82.05 | 80.00
  at Month 12 | 79.55 | 79.49 | 80.00

10. Secondary Outcome: Percentage of Children Without Higher Basal LH and Estradiol or Testosterone
Time Frame: at 2 days after second triptorelin injection (Day 171)
Population: AOC Subset is defined as 50% of the population randomly assigned
Measure: Number; unit: percentage of participants
Groups:
- AOC Subset: All children in AOC subset who received triptorelin 22.5 mg, intramuscular (IM), at Day 1 and Day 169
Arm/Group | AOC Subset
Number analyzed (Participants) | 22
percentage of participants | 13.64

11. Secondary Outcome: Change From Baseline in Height-for-age Z-score Per 2000 CDC Growth Charts at Months 6 and 12
Time Frame: Baseline to Months 6 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Children
Number analyzed (Participants) | 44
Z-score
  at Month 6 | 0.05 (0.20)
  at Month 12 | 0.00 (0.27)

12. Secondary Outcome: Change From Baseline in Height-for-age Percentile Per 2000 CDC Growth Charts at Months 6 and 12
Time Frame: Baseline to Months 6 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | Children
Number analyzed (Participants) | 44
percentile
  at Month 6 | 1.01 (3.21)
  at Month 12 | 0.91 (4.39)

13. Secondary Outcome: Change From Baseline in Growth Velocity at Months 6 and 12
Time Frame: Baseline to Months 6 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Children
Number analyzed (Participants) | 44
cm/year
  at Month 6 | 6.84 (2.33)
  at Month 12 | 6.05 (1.7)

14. Secondary Outcome: Percentage of Participants Without Bone Age / Chronological Age Ratio Increase From Baseline at Months 6 and 12
Time Frame: Baseline to Months 6 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants
  at Month 6 | 63.64
  at Month 12 | 95.45

15. Secondary Outcome: Percentage of Children Achieving Stabilization of Sexual Maturation at Months 6 and 12
Time Frame: at Months 6 and 12
Population: Intention to treat, defined as all participants enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Children
Number analyzed (Participants) | 44
percentage of participants
  at Month 6 | 90.91
  at Month 12 | 88.64

16. Secondary Outcome: Percentage of Girls With Regression of Uterine Length Compared to Baseline at Months 6 and 12
Time Frame: Baseline to Months 6 and 12
Population: Intention to treat girls, defined as all girls enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Girls
Number analyzed (Participants) | 39
percentage of participants
  at Month 6 | 69.23
  at Month 12 | 76.92

17. Secondary Outcome: Percentage of Boys With Absence of Progression of Testis Volumes Compared to Baseline at Months 6 and 12
Time Frame: Baseline to Months 6 and 12
Population: Intention to treat boys, defined as all boys enrolled
Measure: Number; unit: percentage of participants
Arm/Group | Boys
Number analyzed (Participants) | 5
percentage of participants
  at Month 6 | 100.00
  at Month 12 | 100.00

ADVERSE EVENTS:
Arm/Group | Children
Serious Adverse Events (participants affected / at risk) | 1/44
Other Adverse Events (participants affected / at risk) | 20/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children (N=44)
Device related infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children (N=44)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Headache (Nervous system disorders) | 6 (7)
Gastroenteritis (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or scientific communication related to this study can only take place once the agreement between the Sponsor and the Investigator has been reached.